CLINICAL TRIAL: NCT02183116
Title: Open Study to Access the Efficacy and Safety of Meloxicam 7.5mg in Patients With Osteoarthritis of the Knee
Brief Title: A Study to Access the Efficacy and Safety of Meloxicam in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107.228
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Meloxicam

ARMS (1):
- Meloxicam (Experimental)
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Meloxicam
  Other Names: Mobic

SUMMARY:
To Access the Efficacy and Safety of Meloxicam 7.5mg once daily over a treatment period of 56 days

ELIGIBILITY:
Inclusion Criteria:

- Osteoarthritis of the knee requiring the therapy with non-steroidal anti-inflammatory drugs (NSAIDs)

Exclusion Criteria:

none

Ages: 34 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-10; Primary Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on active movement assessed by a 100 mm visual analogue scale (100 mm, VAS) | Baseline, 8 weeks after first drug administration

SECONDARY OUTCOMES:
Change from baseline in Lequesne index | Baseline, 8 weeks after first drug administration
Change from baseline in physical examination (tenderness) | Baseline, 8 weeks after first drug administration
Assessment of significant change from baseline in status according endoscopy | Baseline, 8 weeks after first drug administration
Assessment of significant change from baseline in gastrointestinal (GI) symptoms score | Baseline, 8 weeks after first drug administration
Assessment of significant change from baseline in laboratory values | Baseline, 8 weeks after first drug administration
Number of Patients with Adverse Events | Up to 8 weeks after first drug administration
Assessment of significant change from baseline in physical examination (swelling) | Baseline, 8 weeks after treatment